CLINICAL TRIAL: NCT01159457
Title: Engerix B Versus Sci-B-Vac Immunization in a Celiac Population of Non-responders to Primary Hepatitis B Immunization Series - a Randomized Controlled Trial
Brief Title: Comparison of Engerix B Vaccine Versus Sci-B-Vac Vaccine in Celiac Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Lena Rachman, Shaare Zedek Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 15364.ct.il
Record Dates: First submitted 2010-07-08; First posted 2010-07-09 (Estimated); Last update posted 2011-04-15 (Estimated); Status verified 2011-04

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Hepatitis B vaccination
MeSH Terms: conditions — Celiac Disease

ARMS (2):
- 1 (Active Comparator): celiac patients who did not respond to initial hepatitis B vaccine series , will receive Sci-B-Vac vaccination series
  Interventions: Biological: Hepatitis B vaccination (Sci-B-Vac)
- 2 (Active Comparator): celiac patients who did not respond to initial hepatitis B vaccine series , will receive Engerix 3-dose vaccination series
  Interventions: Biological: Hepatitis B vaccination (EngerixB)

INTERVENTIONS:
Biological: Hepatitis B vaccination (Sci-B-Vac) — A dose of 5mcg (0.5 ml) (up to 10yr old) and 10mcg (1.0 ml)(above 10yr old) of the recombinant HBV vaccine will be administered intramuscularly at zero, one and six months intervals
  Arms: 1
Biological: Hepatitis B vaccination (EngerixB) — A dose of 10mcg (0.5 ml) of the recombinant HBV vaccine will be administered intramuscularly at zero, one and six months intervals
  Other Names: GSK
  Arms: 2

SUMMARY:
Celiac disease and infection with hepatitis B virus (HBV) are very prevalent worldwide and carry a high morbidity rate. It has been recently shown that patients with celiac disease very often fail to develop immunity after standard vaccination for HBV during infancy. In this study, we will evaluate whether a second vaccination series with a different vaccine, Sci-B-Vac, results in a better immunological response in celiac patients. Eligible patients will be randomized to receive a 3-dose vaccination series with Engerix or Sci-B-Vac vaccines.. Rate of responders and level of immunity will be compared. This study will facilitate better protection of celiac patients to this potentially deadly virus.

ELIGIBILITY:
Inclusion Criteria:

* Patients above 1 year of age with confirmed diagnosis of celiac disease by characteristic symptoms, serology and small bowel biopsy.
* Completion of the IM HBV vaccine series in infancy.
* HBsAb titer of <10mIU/mL at the time of enrollment.

Exclusion Criteria:

* Immunocompromised subjects or those receiving medications that may modulate or suppress the immune system (i.e. azathioprine, 6-MP, steroids).
* Inability to obtain written informed consent and patients' assent, as appropriate by the maturity age.

Ages: 1 Year to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 210 (Estimated)
Dates: Start 2011-04; Primary Completion 2012-06 (Estimated); Study Completion 2013-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the geometric mean titers of anti-HBs between the Engerix B group and the Sci-B-Vac group | two years

SECONDARY OUTCOMES:
Rate of responders four weeks after the completion of the series | two years
Rate and characteristics of adverse drug reactions | two years
Numerical increase in the antibodies titer before and after vaccination | two years
Rate of responders in the cross over phase. | two years
Association between the HBsAg-specific cytokine secreting PBMCs by the ELISPOT assay and vaccine response | two years
Association between genetic make-up and vaccine response | two years

CONTACTS AND LOCATIONS:
Overall Officials: Lena Rachman, MD, Principal Investigator — Shaheed Ziaur Rahman Medical College
Locations (1):
- SZMC, Jerusalem, Israel